CLINICAL TRIAL: NCT02584712
Title: Effect of Exercise Training in Autonomic Modulation in Breast Cancer Patients Treated With Doxorubicin
Brief Title: Effect of Exercise Training in Autonomic Modulation in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Maranhao (Other)
Responsible Party: Principal Investigator, Cristiano Teixeira Mostarda, PhD Teacher and Investigator, Federal University of Maranhao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUMaranhao
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Breast Neoplasms; Autonomic Nervous System Diseases
MeSH Terms: conditions — Breast Neoplasms; Autonomic Nervous System Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): This group do not participated in the intervention protocol (exercise training), and was followed throughout the entire process. Autonomic activity was assessed before and after 4 weeks.
- Exercise Training (Active Comparator): This group undergone exercise training intervention during 4 weeks.
  Interventions: Other: Combined Exercise Training

INTERVENTIONS:
Other: Combined Exercise Training — This intervention consisted in 4 weeks of strength, flexibility and aerobic exercises made at the hospital and at home.
  Other Names: Exercise
  Arms: Exercise Training

SUMMARY:
The aim of this study is to evaluate the effect of exercise training in the autonomic nervous system activity in breast cancer patients, who underwent doxorubicin medication.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients at stages 1, 2 and 3;
* Sedentary;
* Currently at treatment;
* 4-6 months after surgery

Exclusion Criteria:

* Musculoskeletal injuries or disorders;
* Mental illnesses
* Stage 4 (Metastasis)
* Enrolled in other exercise program

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction in Low Frequency Heart rate variability component (LF) | 4 weeks
  This reduction is positive, indicating a reduction in sympathetic activity and thus the cardiovascular risk
Increase in High Frequency heart rate variability component (HF) | 4 weeks
  Means a increase in parasympathetic activity, which is correlated to reduction in cardiovascular risk

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano T Mostarda, PhD, Principal Investigator — Federal University of Maranhao